CLINICAL TRIAL: NCT01011075
Title: A Phase II Study of Intermittent Gleevec® (Imatinib Mesylate) and Weekly Paclitaxel in Patients Aged 70 or Older With Advanced Non-small Cell Lung Cancer
Brief Title: Study of Gleevec and Weekly Paclitaxel in Patients Aged 70 or Older With Advanced Non-small Cell Lung Cancer
Acronym: 6137p
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST CST1571BUS240; NCI-2011-02947 (Registry Identifier: NCI Clinical Trials Reporting Program); 6137p (Other: Novartis)
Record Dates: First submitted 2009-10-14; First posted 2009-11-11 (Estimated); Results first posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung cancer,; Non-small cell lung cancer; NSCLC; Metastatic; Gleevec; elderly
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasm Metastasis | interventions — Imatinib Mesylate; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imatinib mesylate + Paclitaxel (Experimental): Paclitaxel 90 mg/m2 IV on days 3, 10, 17 Imatinib (Gleevec) 600 mg/day, oral administration in 4-day pulses bracketing each paclitaxel infusion (days 1-4; 8-11; 15-18) Cycle length: 28 days Number of cycles: up to 6
  Interventions: Drug: Imatinib mesylate; Drug: Paclitaxel

INTERVENTIONS:
Drug: Imatinib mesylate — Imatinib (Gleevec) 600 mg/day, oral administration in 4-day pulses(days 1-4; 8-11; 15-18) Cycle length: 28 days Number of cycles: up to 6
  Other Names: Gleevec
Drug: Paclitaxel — Paclitaxel 90 mg/m2 IV on days 3, 10, 17 Cycle length: 28 days Number of cycles: up to 6
  Other Names: Taxol

SUMMARY:
This study will evaluate the clinical efficacy of combining Gleevec (imatinib mesylate), a PDGFR antagonist, with front-line, single-agent paclitaxel in a cohort of elderly patients with advanced, non-small cell lung cancer.

DETAILED DESCRIPTION:
Paclitaxel 90 mg/m2 IV on days 3, 10, 17 Imatinib 600 mg/day, oral administration in 4-day pulses bracketing each paclitaxel infusion (days 1-4; 8-11; 15-18) Cycle length: 28 days Number of cycles: up to 6

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Histologic or cytologic diagnosis of non-small cell lung cancer
* At least one site of measurable disease, as defined by the modified RECIST criteria (See section 7.6)
* Stage IIIB with pleural effusion or Stage IV disease. Includes patients who received surgery alone for early stage disease, now in relapse with advanced disease. Staging is according to the American Joint Committee on Cancer classification scheme, 6th edition.48
* Adequate hepatic, renal and marrow function

  * Liver function tests: total bilirubin < 1.25 x upper limit of normal (ULN), AST and ALT < 2.5 x ULN, Creatinine < 1.5 x ULN
  * Baseline absolute neutrophil count > 1500/μL
  * Baseline platelet count > 100,000/μL
* ECOG Performance Status 0, 1 or 2 at the time of informed consent. (See Appendix 1)
* Written, voluntary consent
* Patients with reproductive potential must use an acceptable contraceptive method. Such methods include: 1) Male hormonal contraception; 2) Partner without reproductive potential, including post-menopausal status or history of tubal ligation; 3) Partner with intrauterine device (IUD) or contraceptive vaginal ring; 4) Partner takes oral contraceptive pill, wears contraceptive patch, or has contraceptive implant; 5) Routine use of barrier method, such as condoms or diaphragm, during sexual intercourse.

Exclusion Criteria:

Uncontrolled brain metastasis. Patients with known brain metastasis must have completed treatment with surgery, radiation or both. In addition, they must be off corticosteroids.

* Symptomatic neuropathy (Grade 2 or higher)
* Prior chemotherapy for advanced non-small cell lung cancer. (Prior adjuvant, neoadjuvant, or chemoradiotherapy for NSCLC is permitted, provided at least 6 months elapsed prior to documented metastatic recurrence.)
* Patient is < 5 years free of another primary malignancy, except: a) if the other malignancy is basal cell carcinoma or cervical carcinoma in situ or b) if the other primary malignancy is not considered clinically significant and is requiring no active intervention
* Prior radiation therapy to > 25% of bone marrow
* Grade III/IV congestive heart failure, as defined by NYHA criteria, or myocardial infarction within 6 months.
* Any serious or uncontrolled concomitant disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* Patient has known chronic liver disease, e.g. diagnosis of chronic active hepatitis or cirrhosis.
* Major surgery two weeks prior to study treatment
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent
* Any condition requiring continuous administration of systemic corticosteroids.
* The patient is on therapeutic anti-coagulation with warfarin.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bauman, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (3):
- United States (3):
  - University of New Mexico Cancer Center @ Lovelace Medical Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Univ. of Washington Fred Hutchinson Cancer Research Center (UW-FHCRC), Seattle, Washington

REFERENCES:
- [Result] Bauman JE, Eaton KD, Wallace SG, Carr LL, Lee SJ, Jones DV, Arias-Pulido H, Cerilli LA, Martins RG. A Phase II study of pulse dose imatinib mesylate and weekly paclitaxel in patients aged 70 and over with advanced non-small cell lung cancer. BMC Cancer. 2012 Oct 3;12:449. doi: 10.1186/1471-2407-12-449. PMID 23033932

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject screening for this study began effective 08/12/2009 at the UNM Cancer Center. Recruitment was conducted through the outpatient clinic. Patients were recruited until 04/30/2010.
Groups:
- Imatinib Mesylate and Paclitaxel: Experimental: Treatment (enzyme inhibitor, chemotherapy) Patients receive paclitaxel IV on days 3, 10, and 17 and imatinib mesylate PO QD on days 1-4, 8-11, and 15-18. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Imatinib Mesylate and Paclitaxel
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate and Paclitaxel
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.5 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rates according to RECIST criteria (version 1.0) expressed as percentage of evaluable patients.
Time Frame: 6 months
Population: 6 of the enrolled 34 patients were inevaluable for the primary endpoint of Response Rate due to withdrawal or death prior to first response assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Imatinib Mesylate and Paclitaxel
Number analyzed (Participants) | 28
Percentage of Participants | 32 [17.4 to 50.5]

2. Secondary Outcome: Overall Survival
Description: Overall survival as measured by the Kaplan-Meier method
Time Frame: 12 Months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib Mesylate and Paclitaxel
Number analyzed (Participants) | 28
Months | 7.3 [5 to 16]

3. Secondary Outcome: Progression Free Survival
Description: Number of months post treatment without measurable progression according to RECIST criteria (version 1.0)
Time Frame: 12 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib Mesylate and Paclitaxel
Number analyzed (Participants) | 28
Months | 3.6 [3 to 7]

4. Secondary Outcome: Toxicities
Description: Adverse events of grade 3 or higher, according to CTCAE version 3
Time Frame: 12 months
Population: All enrolled and treated patients were evaluated for grade 3 or higher toxicities.
Measure: Number; unit: Number of events
Arm/Group | Imatinib Mesylate and Paclitaxel
Number analyzed (Participants) | 34
Number of events | 34

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Imatinib Mesylate and Paclitaxel
Serious Adverse Events (participants affected / at risk) | 4/34
Other Adverse Events (participants affected / at risk) | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate and Paclitaxel (N=34)
Cardiac arrest (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate and Paclitaxel (N=34)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Systolic dysfunction (Cardiac disorders) | 2
Edema (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 10
Infection (Infections and infestations) | 4
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Bladder/Kidney stone (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days